CLINICAL TRIAL: NCT02034201
Title: Clinical Efficacy of Lisdexamfetamine for Methamphetamine Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 119273; R21DA034824-01A1 (NIH)
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Methamphetamine Dependence
MeSH Terms: interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Lisdexamfetamine (Active Comparator): Lisdexamfetamine will be admistered at 140 mg orally daily through week 6 of the protocol.
  Interventions: Drug: Lisdexamfetamine
- Placebo (Placebo Comparator): Placebo will be administered orally daily through week 6 of the protocol.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine
  Arms: Lisdexamfetamine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Methamphetamine dependence is a serious public health problem, with methamphetamine abusers being at risk for significant morbidity and mortality, including HIV. To date, no medication or psychotherapeutic strategy has shown robust, long-term efficacy in treating this disorder. This clinical trial will examine whether lisdexamfetamine shows promise in alleviating withdrawal symptoms and preventing relapse relative to placebo in recently-abstinent methamphetamine dependent individuals. Findings of this study will not only shed light on whether lisdexamfetamine may improve upon treatment for this disorder but also inform future medication development strategies for improving treatment for drug dependence disorders. Discovering efficacious limited risk interventions that show more robust, longer-term outcomes would be beneficial both to the individual and society.

ELIGIBILITY:
Inclusion Criteria:

1. Age (18-65 yrs).
2. Participants must fulfill DSM-IV criteria for Methamphetamine dependence These criteria will be ascertained in the following manner: the physician will determine whether the individual is appropriate based on clinical assessments and the patient will also need to meet criteria for methamphetamine dependence based on administration of the SCID.
3. Self-reported average METH use of at least 250 mg of methamphetamine per occasion at least once weekly during the preceding 3-month period.
4. A positive urine toxicology screen for methamphetamine. Participants must submit a urine sample negative for drugs of abuse (opiates, benzodiazepines, cocaine and PCP) other than methamphetamine or marijuana during the week prior to starting the study.
5. Women of child-bearing potential will be included provided they 1) have a negative pregnancy test, 2) agree to adequate contraception (tubal ligation, hysterectomy, barrier contraceptive method or oral contraceptive method) to prevent pregnancy during the study and 3) are not nursing.
6. Normal blood pressure with SBP >89 and < 141, DBP >59 and < 91.

Exclusion Criteria:

1. Current suicidality or psychosis
2. Current cocaine dependence or opioid, alcohol, or sedative physical dependence
3. Major hepatic or cardiovascular disorder (including history of myocardial infarction, cardiovascular disease, or history of or currently clinically significant ECG abnormality) or unstable medical condition that contraindicates study participation
4. History of schizophrenia or bipolar type I disorder
5. Use of medications that would be expected to have major interaction with LDX including psychotropics
6. Medical contraindication to receiving LDX
7. Positive drug screen for cocaine, opiates, sedatives or PCP.
8. History of Seizure disorder
9. Documented hypersensitivity to sympathomimetic amines
10. LFT >3xULN
11. Pregnancy/nursing
12. Current use or past 2 weeks use of MAOi
13. History of Narrow-angle glaucoma

g.n. History of Hyperthyroidism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-02; Primary Completion 2016-05-19 (Actual); Study Completion 2016-05-19 (Actual)

PRIMARY OUTCOMES:
Percentage of participants that relapse to methamphetamine use. | 9 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States